CLINICAL TRIAL: NCT07022665
Title: Influence of Hospital Volume on Mortality and Short-term Postoperative Outcomes in Uncomplex General Surgery in Switzerland: A Retrospective National Registry Study
Brief Title: Influence of Hospital Volume on Mortality and Short-term Postoperative Outcomes in Uncomplex General Surgery in Switzerland
Status: Completed | Type: Observational
Sponsor: Cantonal Hospital of St. Gallen (Other)
Responsible Party: Principal Investigator, Yanic Ammann, Principal Investigator, Cantonal Hospital of St. Gallen
Other Study IDs: hospital volume surgery
Record Dates: First submitted 2025-05-26; First posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Cholecystolithiasis; Cholecystitis; Inguinal Hernia; Femoral Hernia; Umbilical Hernia; Appendicitis
MeSH Terms: conditions — Cholecystolithiasis; Cholecystitis; Hernia, Inguinal; Hernia, Femoral; Hernia, Umbilical; Appendicitis | interventions — Appendectomy; Cholecystectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Appendicectomy
  Interventions: Procedure: Appendicectomy
- Cholecystectomy
  Interventions: Procedure: Cholecystectomy
- Umbilical hernia repair
  Interventions: Procedure: Umbilical hernia repair
- Inguinal and/or femoral hernia repair
  Interventions: Procedure: Inguinal and/or femoral hernia repair

INTERVENTIONS:
Procedure: Appendicectomy — Appendicectomy for appendicitis
  Groups: Appendicectomy
Procedure: Cholecystectomy — Cholecystectomy for cholecystolithiasis and/or cholecystitis
  Groups: Cholecystectomy
Procedure: Umbilical hernia repair — Any kind of umbilical hernia repair
  Groups: Umbilical hernia repair
Procedure: Inguinal and/or femoral hernia repair — Any kind of inguinal and/or femoral hernia repair
  Groups: Inguinal and/or femoral hernia repair

SUMMARY:
The effect of centralisation measures on the operative outcomes after any type of surgery in Switzerland has not been highlighted yet. This study aims to investigate the influence of the annual case-specific hospital volume on uncomplex general surgery. The four operations investigated are appendectomy, cholecystectomy, umbilical hernia repair, and inguinal/femoral hernia repair.

ELIGIBILITY:
Inclusion Criteria:

* All patients with appendicectomy for appendicitis, cholecystectomy for cholecystolithiasis and/or cholecystitis , umbilical hernia repair, or inguinal and/or femoral hernia repair

Exclusion Criteria:

* incomplete case documentation
* age under 20 years
* other hospitals than general or surgical hospitals
* no index operation

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients with with appendicectomy for appendicitis, cholecystectomy for cholecystolithiasis and/or cholecystitis , umbilical hernia repair, or inguinal and/or femoral hernia repair operated in Switzerland between 2013 and 2022.
Sampling Method: Non-Probability Sample
Enrollment: 399701 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Mortality | Periprocedural
  The association between the hospital volume and the postoperative mortality Mortality Yes or No Hospital volume as marginal effect Association with GAM logistic regression

SECONDARY OUTCOMES:
Reoperation | Periprocedural
  The association between the hospital volume and the reoperation rate Reoperation Yes or No Hospital volume as marginal effect Association with GAM logistic regression
Length of hospital stay | Periprocedural
  The association between the hospital volume and the length of hospital stay Length of hospital stay in days Hospital volume as marginal effect Association with quantile regression
Sociodemographic trends | 2013 - 2022

CONTACTS AND LOCATIONS:
Locations (1):
- HOCH Health Ostschweiz, Kantonsspital St.Gallen, Sankt Gallen, St.Gallen, Switzerland

IPD SHARING:
Plan to Share IPD: No